CLINICAL TRIAL: NCT07219615
Title: A PHASE 2B RANDOMIZED, DOUBLE-BLIND, 12-WEEK PLACEBO-CONTROLLED STUDY WITH A 12-WEEK DOUBLE-BLIND EXTENSION PERIOD TO EVALUATE THE EFFICACY, SAFETY AND TOLERABILITY OF RITLECITINIB (PF-06651600) IN ADULT PARTICIPANTS WITH CHRONIC SPONTANEOUS URTICARIA
Brief Title: A Study to Learn About Ritlecitinib for the Potential Treatment of Chronic Spontaneous Urticaria in Adults.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981118; 2025-522642-44-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Hives; CSU; Urticaria; Chronic Hives; Itch
MeSH Terms: conditions — Chronic Urticaria; Urticaria; Pruritus | interventions — PF-06651600

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Randomized to Ritlecitinib 50 mg for 24 weeks Periods A and B). In addition to the active Ritlecitinib 50 mg capsule, a placebo matching the Ritlecitinib 100 mg capsule will be given to maintain blind
  Interventions: Drug: Ritlecitinib 50 mg; Drug: Placebo - 100 mg
- Arm 2 (Experimental): Randomized to Ritlecitinib 100 mg for 24 weeks (Periods A and B). In addition to the active Ritlecitinib 100 mg capsule, a placebo matching the Ritlecitinib 50 mg capsule will be given to maintain blind
  Interventions: Drug: Ritlecitinib 100 mg; Drug: Placebo - 50 mg
- Arm 3 (Placebo Comparator): Randomized to placebos matching the Ritlecitinib 50 mg and Ritlecitinib 100 mg capsules will be given to maintain blind from Day 1 to Week 12 (Period A). From Week 12 to Week 24 (Period B), will be switched to Ritlecitinib 100 mg. In addition to the active Ritlecitinib 100 mg capsule, a placebo matching the Ritlecitinib 50 mg capsule will be given to maintain blind.
  Interventions: Drug: Ritlecitinib 100 mg; Drug: Placebo - 50 mg; Drug: Placebo - 100 mg

INTERVENTIONS:
Drug: Ritlecitinib 50 mg — 50 mg Capsule
  Other Names: PF-06651600; Litfulo
  Arms: Arm 1
Drug: Ritlecitinib 100 mg — 100 mg Capsule
  Other Names: PF-06651600; Litfulo
  Arms: Arm 2; Arm 3
Drug: Placebo - 50 mg — Matching Capsule
  Arms: Arm 2; Arm 3
Drug: Placebo - 100 mg — Matching Capsule
  Arms: Arm 1; Arm 3

SUMMARY:
The purpose of the study is to learn about the safety and effects of the study medicine (called ritlecitinib) for the treatment of chronic spontaneous urticaria (CSU) that is not effectively treated by antihistamines which are used to stop the body's "allergy alarm system" from overreacting. Chronic spontaneous urticaria is a disease that causes itchy hives and swellings in the deep layers of skin and fatty tissue just underneath the skin that come and go without a clear reason.

This study will look at both the 50 milligrams (mg) once daily (QD) oral dose and 100 milligrams (mg) once daily (QD) oral dose and compare them to placebo (pill with no active medicine).

This study is seeking participants who:

* Are 18 years of age or older
* Have a diagnosis of chronic spontaneous urticaria for 3 months or more that has not been controlled well with antihistamine treatment.
* Do not have any other skin conditions associated with chronic itching or itching caused mainly by known triggers.
* Are willing to stop all other treatments that they may be taking for chronic spontaneous urticaria other than a second-generation antihistamine (sgAH).

About 150 participants will take part in this study. Participants will be chosen by chance, like drawing names out of a hat, to receive either the 50 mg dose or 100 mg dose or placebo, taken by mouth once daily for 12 weeks( Period A). Thereafter the participants on 50 mg and 100 mg will continue on their doses while the participants receiving placebo will be switched to 100mg for an additional 12 weeks (Period B). The 2 doses of ritlecitinib in this study will be compared to each other and to the placebo. This will help to see if the 50 mg and/or 100 mg dose of ritlecitinib is safe and effective.

Participants will be in this study for about 8 months. During the study, participants will need to visit the study site up to 9 times. Participants will undergo various tests and procedures such as:

* Physical examinations,
* Hearing tests,
* Blood tests,
* X-ray,
* ECG (electrocardiogram),
* Participants will also be asked to complete questionnaires every day about their chronic spontaneous urticaria in an electronic diary.

ELIGIBILITY:
Inclusion Criteria:

Age:

1. 18 years of age or older (or the minimum legal adult age as defined per local regulations, whichever is greater) at screening.

   Disease Characteristics:
2. Participants must meet the following Chronic Spontaneous Urticaria (CSU) criteria:

   a. Chronic spontaneous urticaria diagnosis for ≥3 months at the time of screening (with the onset date assessed by the Investigator based on all available records) b. Diagnosis of CSU inadequately controlled by second generation antihistamine (sgAH) at the time of randomization, defined as: (i) The presence of itch and hives for ≥6 consecutive weeks prior to screening despite the use of sgAH during this time period.

(ii) Participants must have been on a sgAH at locally approved dose or higher for treatment of CSU for at least 7 consecutive days before screening assessment of UAS7 and ISS7 is initiated.

(iii) Urticaria Activity Score 7 (UAS7) ≥16 (range 0-42) and an Itch Severity Score 7 (ISS7) ≥8 (range: 0-21) during the 7 days prior to randomization Day 1 c. Participants must complete at least 5 Urticaria Activity Score (UAS) eDiary entries during the 7 days immediately preceding randomization (Day 1) to confirm eligibility. If this requirement is not met due to documented, limited circumstances such as technical issues or short-term illness, the screening period may be extended only for the number of days necessary to allow completion of 5 UAS entries within any 7-day window. This extension period must not exceed 7 days.

d. Anti-Immunoglobulin E-naïve (IgE-naïve) and Anti-Immunoglobulin E-experienced (Anti-IgE-experienced) participants. Anti-IgE-experienced participants are defined as meeting any of the following criteria confirmed by the Site Investigator: (i) Did not adequately respond to the approved dosage of an anti-IgE therapy (eg, omalizumab 300 mg Q4W or an alternate approved anti-IgE therapy) for at least 3 months, as assessed by the Investigator (ii) Could not tolerate an anti-IgE therapy (iii) Stopped an anti-IgE therapy for any reason, eg, loss of access e. Anti-IgE-experienced participants must have stopped anti-IgE therapy for at least 16 weeks, or 5 half-lives, whichever is longer, prior to randomization Day 1

Exclusion Criteria:

Medical Conditions:

1. Medical conditions pertaining to CSU and other diseases/conditions affecting the skin

   * Urticaria is solely due to inducible urticaria.
   * Active dermatologic diseases (or conditions) other than chronic urticaria, with urticaria wheals or angioedema symptoms, including but not limited to urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to Complement 1 (C1) inhibitor deficiency).
   * Any other active skin disease associated with chronic itching that might influence, in the investigator's opinion, the study evaluations and results (eg, atopic dermatitis, bullous pemphigold, dermatitis herpetiformis, senile pruritus, etc.).
2. History of severe allergic or anaphylactoid reaction to any kinase inhibitor or a known allergy/hypersensitivity to any component (including excipients) of the study intervention.
3. General Infection History:

   * Having a history of systemic infection requiring hospitalization or parenteral therapy (antimicrobial, antiviral, antiparasitic, antiprotozoal, or antifungal), or as otherwise judged clinically significant by the investigator, within 3 months prior to Day 1.
   * Have active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 1.
   * Evidence or history of untreated, currently treated or inadequately treated active or latent infection with Mycobacterium tuberculosis.
4. Specific Viral Infection History

   * History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
   * Infected with hepatitis B or hepatitis C viruses: all participants will undergo screening for hepatitis B and C for eligibility.
   * Have a known immunodeficiency disorder (including positive serology for HIV at screening) or a first-degree relative with a hereditary immunodeficiency (unless known negative carrier status).
5. Other Medical Conditions

   * Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (eg, untreated hyperthyroidism or hypothyroidism), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator or Pfizer (or designee), the participant is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle requirements.
   * Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating, or progressive.
   * Abnormal findings on the screening chest imaging (eg, chest x-ray) including, but not limited to, presence of active TB or other infections, cardiomyopathy, or malignancy. Chest imaging may be performed up to 12 weeks prior to Screening.
   * Have any malignancies or have a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
   * Have a history of any lymphoproliferative disorder such as Epstein-Barr Virus (EBV)-related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
   * Significant trauma or major surgery within 1 month of the first dose of study drug or considered in imminent need for surgery. Participants with elective surgery scheduled to occur during the study can only be enrolled with approval of the sponsor.
6. Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study. Any psychiatric condition including recent or active suicidal ideation or behavior that protocol-defined criteria.

   Prior/Concomitant Therapy:
7. Current or prior use of any prohibited medication(s), vaccine(s), or treatment(s) within the protocol defined timelines.

   Prior/Concurrent Clinical Study Experience:
8. Previous administration of an investigational product (drug or vaccine) within 8 weeks or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during participation in this study.

   Diagnostic Assessments:
9. Any exclusionary abnormalities in laboratory values at Screening, as assessed by the study-specific laboratory and, if deemed necessary, confirmed by a single repeat.
10. Screening standard 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.

    Other Exclusion Criteria:
11. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Urticaria Activity Score 7 (UAS7) at Week 12 | Week 12
Incidence of Treatment Emergent Adverse Events, Serious Adverse Events, and Adverse Events leading to discontinuation | Week 12

SECONDARY OUTCOMES:
Change from baseline in UAS7 at all timepoints except Week 12 | Week 1 through Week 11
Change from baseline in Itch Severity Score 7 (ISS7) at Week 12 | Week 12
Change from baseline in Hives Severity Score 7 (HSS7) at Week 12 | Week 12
Achieving complete response defined as UAS7=0 at Week 12 | Week 12
Achieving UAS7 ≤6 at Week 12 | Week 12
Achieving complete response defined as ISS7=0 at Week 12 | Week 12
Achieving complete response defined as HSS7=0 at Week 12 | Week 12
Time to achieving UAS7 ≤6 | Week 12
Time to achieving improvement from baseline ≥10 in UAS7 | Week 12
Incidence of TEAEs, SAEs, and AEs leading to discontinuation | After Week 12 through Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Revival Research Institute, LLC, Troy, Michigan
  - Allergy, Asthma and Clinical Research, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981118